CLINICAL TRIAL: NCT05958355
Title: Effects of Functional Postural Control Training on Functional Performance in People With Parkinson's Disease With Freezing of Gait
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Ray-Yau Wang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NYCU112071AF
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Parkinson Disease
Keywords: Freezing of gait; Functional postural control training; Functional performance; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional postural control training (Experimental): The training includes (1) Maintaining a stationary posture in a standing position for a total of 10 minutes, (2) Posture control training involving unilateral lower limb stepping movements for a total of 10 minutes, and (3) Advanced walking task training, including sudden stops, turns, ball raises, and obstacle crossing during walking, for a total of 10 minutes.
  Interventions: Other: Functional postural control training
- Treadmill training (Active Comparator): The subjects in the control group performed a 30-minute walking session on a treadmill at a self-selected speed.
  Interventions: Other: Treadmill training

INTERVENTIONS:
Other: Functional postural control training — All participants will receive functional postural control training for 30 minutes/ session, 3 sessions/ weeks, for 4 weeks (a total of 12 training sessions).
  Arms: Functional postural control training
Other: Treadmill training — All participants will receive treadmill training for 30 minutes/ session, 3 sessions/ weeks, for 4 weeks (a total of 12 training sessions).
  Arms: Treadmill training

SUMMARY:
The purpose of this single-blinded, randomized controlled study aims to establish the effects of functional postural control training on functional performance and FOG in PD individuals with FoG as compared with treadmill training.

DETAILED DESCRIPTION:
Background and purpose: Freezing of gait (FoG), is a common sign in patients with Parkinson's disease (PD), especially at the advanced stage. Advanced functional activities, such as dual task walking, turning, or crossing a door often induce the FOG. FoG is a complex phenomenon which pathophysiology is currently unknown. However, previous studies have found that postural instability may be a risk factor for FoG. In addition, previous studies have suggested the interactions between FoG and postural instability. Treadmill training has been shown to be relatively more effective to improve FoG than other interventions. On the other hand, postural control training was demonstrated to improve the severity of FoG and postural control in freezers. However, no study has investigated the effectiveness of functional postural control training on functional performance and FOG. Therefore, this study aims to establish the effects of functional postural control training on functional performance and FOG in PD individuals with FoG as compared with treadmill training.

Methods: This study is a single-blinded randomized controlled trial. Twenty PD people with FoG will be recruited and randomized to the experimental and control group. The experimental group will receive functional postural control training, and the control group will receive treadmill training. Each intervention is 30 minutes/ session, 3 sessions/ weeks, for 4 weeks. The primary outcome is functional performance, which will measure the walking speed, cadence, and step length in the four conditions, including (1) Time up and go test, (2) Dual task Time up and go test, (3) 360º turning in place, and (4) Walking through the door. The secondary outcome is the severity of FoG which is assessed by the New Freezing of Gait Questionnaire (NFOGQ). All outcomes will be assessed before and after the training program. Demographic data at baseline will be analyzed by using Chi-square test or independent T-test. Two-way repeated ANOVA will be performed to analyze the primary and secondary outcomes. The significance level is set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Hoehn and Yahr stage 2~4
* Age between 50 to 80 years
* New Freezing of Gait Questionnaire score > 1
* Able to walk independently for at least 10 meters
* MMSE score ≥24

Exclusion Criteria:

* Neurological diseases other than PD
* Any cardiovascular, pulmonary, or orthopedic conditions that would impact participation in the study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Functional performance-Time up and go test-speed(m/s) | Change from baseline time up and go test walking speed and up to 4 weeks (pre- and post-test)
  Using GaitUp system to evaluate walking speed during the Time Up and Go test.
Functional performance-Time up and go test-cadence (steps/ min) | Change from baseline time up and go test cadence and up to 4 weeks (pre- and post-test)
  Using GaitUp system to evaluate cadence during the Time Up and Go test.
Functional performance-Time up and go test-step length (m) | Change from baseline time up and go test step length and up to 4 weeks (pre- and post-test)
  Using GaitUp system to evaluate step length during the Time Up and Go test.
Functional performance-dual task Time up and go test-speed(m/s) | Change from baseline dual task time up and go test walking speed and up to 4 weeks (pre- and post-test)
  Using GaitUp system to evaluate walking speed during the dual task Time up and go test.
Functional performance-dual task Time up and go test-cadence (steps/ min) | Change from baseline dual task time up and go test cadence and up to 4 weeks (pre- and post-test)
  Using GaitUp system to evaluate cadence during the dual task Time up and go test.
Functional performance-dual task Time up and go test-step length (m) | Change from baseline dual task time up and go test step length and up to 4 weeks (pre- and post-test)
  Using GaitUp system to evaluate step length during the dual task Time up and go test.
Functional performance-360º turning in place-speed(m/s) | Change from baseline 360º turning in place speed and up to 4 weeks (pre- and post-test)
  Using GaitUp system to evaluate speed during the 360º turning in place test.
Functional performance-360º turning in place-cadence (steps/ min) | Change from baseline 360º turning in place cadence and up to 4 weeks (pre- and post-test)
  Using GaitUp system to evaluate cadence during the 360º turning in place test.
Functional performance-360º turning in place-step length (m) | Change from baseline 360º turning in place step length and up to 4 weeks (pre- and post-test)
  Using GaitUp system to evaluate step length during the 360º turning in place test.
Functional performance-Walking through the door-speed(m/s) | Change from baseline walking through the door speed and up to 4 weeks (pre- and post-test)
  Using GAITRite® system to evaluate walking speed during walks through the door.
Functional performance-Walking through the door-cadence (steps/ min) | Change from baseline walking through the door cadence and up to 4 weeks (pre- and post-test)
  Using GAITRite® system to evaluate cadence during walks through the door.
Functional performance-Walking through the door-step length (m) | Change from baseline walking through the door step length and up to 4 weeks (pre- and post-test)
  Using GAITRite® system to evaluate step length during walks through the door.

SECONDARY OUTCOMES:
New Freezing of Gait Questionnaire (NFOGQ) | Change from baseline New Freezing of Gait Questionnaire and up to 4 weeks (pre- and post-test)
  Use the New Freezing of Gait Questionnaire (NFOGQ)-Chinese version to assess the severity of freezing of gait.
  The score ranged from 0 to 29. Higher scores show increased severity in freezing of gait.

CONTACTS AND LOCATIONS:
Overall Officials: Ray-Yau Wang, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan